CLINICAL TRIAL: NCT07164469
Title: Phase 2 Trial of CD70.CAR NK Cells for Patients With Primary Refractory or Early Relapsed Diffuse Large B-Cell Lymphoma and Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0986; NCI-2025-06569 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-09-04; First posted 2025-09-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1st Dose: Treatment with Rimiducid + CD70.CAR NK Cells for Patients with DLBCL and HL (Experimental): Patients will receive lymphodepleting chemotherapy with fludarabine and cyclophosphamide from days -5 to -3, prior to infusion of CD70.CAR NK cells on day 0, on an outpatient or inpatient as clinically indicated.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: CD70.CAR NK Cells; Drug: Rimiducid (AP1903)
- 2nd Dose: Treatment with Rimiducid + CD70.CAR NK Cells for Patients with DLBCL and HL (Experimental): Patients will receive lymphodepleting chemotherapy with fludarabine and cyclophosphamide from days -5 to -3, prior to infusion of CD70.CAR NK cells on day 0, on an outpatient or inpatient as clinically indicated.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: CD70.CAR NK Cells; Drug: Rimiducid (AP1903)

INTERVENTIONS:
Drug: Fludarabine — Given by IV
  Other Names: Fludara
Drug: Cyclophosphamide — Given by IV
  Other Names: Cytoxan; Neosar
Drug: CD70.CAR NK Cells — Given by IV Infusion
Drug: Rimiducid (AP1903) — Given by IV Infusion

SUMMARY:
This clinical research study is to learn if CD70.CAR NK cell therapy can help to control early relapsed or primary refractory DLBCL and cHL.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of the study is to determine the efficacy of CB-derived CD70.CAR NK cell therapy in patients with primary refractory or early relapsed DLBCL and HL, as determined by the 2-year event-free survival rate.

Secondary Objectives:

* To determine the antitumor activity pf CB-derived CD70.CAR NK cells, as determined by the response rate (ORR) and complete response (CR) rate.
* To establish the safety of this treatment.
* To quantify the persistence of infused CB-derived CD70.CAR NK cells in the peripheral blood.
* To conduct comprehensive immune studies by evaluating tissue and blood-based biomarkers associated with response and resistance to CD70.CAR NK cells.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age.
2. Diagnosis of cHL or DLBCL that is either:

   * Primary refractory, defined as not having achieved a CR with frontline therapy or having relapsed within 3 months.
   * Early relapsed (≤ 12 months) after achieving a CR to frontline therapy.
3. Tumor biopsy positive for CD70 >/= 10% by immunohistochemistry or flow cytometry.
4. Measurable disease, defined by one or more histologically confirmed hypermetabolic lesion on PET/CT scan.
5. ECOG PS ≤ 2 (Karnofsky ≥60%).
6. Adequate blood counts (WBC > 2K, HGB > 8 g/dL, platelets > 50K).
7. Creatinine clearance ≥ 30 ml/min.
8. ALT and/or AST ≤ 3 x ULN, and bilirubin and ALP ≤ 2 x ULN.
9. FEV1, FVC and DLCOc ≥ 50%.
10. LVEF ≥40%, without active arrythmias.
11. If female of child-bearing potential, she must not be pregnant or breastfeeding and is required to have a negative urine or serum pregnancy test prior to enrollment.
12. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
13. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
14. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
15. Patients with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
16. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.

    To be eligible for this trial, patients should be class 2B or better.
17. The effects of CAR-NK cells on the developing human fetus are unknown. For this reason and because fludarabine and cyclophosphamide, as well as other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114).

    * This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following: Postmenopausal (no menses in greater than or equal to 12 consecutive months). History of hysterectomy or bilateral salpingo-oophorectomy. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy). History of bilateral tubal ligation or another surgical sterilization procedure.
    * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
    * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CAR NK cell administration.
18. Ability to understand and the willingness to sign a written informed consent document.
19. Agree to sign consent to the long-term follow-up protocol PA17-0843 to fulfill the institutional responsibilities to various regulatory agencies.

Exclusion Criteria:

1. Lymphoma in CR with no measurable sites of disease.
2. Major surgery <4 weeks prior to first dose of study drug.
3. Any other severe or uncontrolled disease or condition which might increase the risk associated with study participation.
4. Any other malignancy known to be active, with the exception of treated cervical intra-epithelial neoplasia and non-melanoma skin cancer.
5. Grade >/= 3 non-hematologic toxicity from prior therapy that has not improved to grade </= 2.
6. Active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA

   >/=10,000 copies/mL, or >/=2,000 IU/mL), or hepatitis C (detectable viral load by HCV RNA PCR).
7. Active infection requiring parenteral antibiotics.
8. HIV infection.
9. Treatment within prior 2 weeks with any anti-cancer agent, investigational or approved.
10. Active central nervous system (CNS) involvement (untreatedparenchymal brain metastasis or positive cytology of cerebrospinal fluid).
11. Life expectancy </= 6 months.
12. Active and uncontrolled neurological disorder.
13. Patients receiving systemic steroid therapy at time of enrollment (physiological replacement doses are allowed) or have received antithymocyte globulin or lymphocyte immune globulin within 14 days of enrollment or alemtuzumab within 28 days of enrollment.
14. Patients receiving immunosuppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2031-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org